CLINICAL TRIAL: NCT03861065
Title: Secondary Versus Tertiary Wound Closure in High Risk Gynecologic Abdominal Surgical Incisions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00055298; NCI-2019-01292 (Other: National Cancer Institute); P30CA012197 (NIH); CCCWFU04418 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Surgical Incision
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tertiary Wound Closure (Experimental): In the alternative tertiary wound closure, the wound will be partially closed rather than being left open. Sutures in the skin will be placed but not closed. A vacuum assisted closure device will be placed over the wound to help healing. After 4-7 days, the vacuum device will be removed, and the participant's doctor will close the wound.
  Interventions: Procedure: Tertiary Wound Closure
- Historical Wound Closure (Active Comparator): The standard approach to your wound would be to leave it partially open and let it heal over a period of 3-6 months ("secondary closure").
  Interventions: Procedure: Historical Wound Closure

INTERVENTIONS:
Procedure: Tertiary Wound Closure — The wound will be closed with what is considered tertiary wound closure. This means, rather than leaving the wound open, the wound will be partially closed after surgery, and then completely closed 4-7 days after surgery.
  Arms: Tertiary Wound Closure
Procedure: Historical Wound Closure — Participants wounds are left partially open to heal.
  Arms: Historical Wound Closure

SUMMARY:
The purpose of this research study is to determine if closing a surgical wound differently is better than the procedure that is currently used. The wound will be closed with what is considered "tertiary intent." This means, rather than leaving the wound open, the wound will be partially closed after surgery, and then completely closed 4-7 days after surgery. The investigators also want to see how this new wound closure process affects your quality of life.

DETAILED DESCRIPTION:
Primary Objective

To compare the percentage of patients whose wound remained closed on postoperative day #30 after tertiary closure compared to historical controls who underwent secondary would closure. We are primarily looking at time to wound closure. We will be able to abstract this information from the postoperative clinic visit notes from patients in the "historical control" cohort. We will identify 20 patients with characteristics described in the inclusion criteria of this study who underwent laparotomy with secondary would closure during the calendar year 2018.

Secondary Objectives

To compare the proportion of acute and chronic wound infection in wounds closed with a tertiary closure technique to historical controls receiving a secondary wound closure.

To compare the length of stay of patients receiving a tertiary wound closure to historical controls receiving a secondary wound closure.

To describe the number of patients receiving a tertiary wound closure that return within 30 days of surgery as compared to historical controls receiving a secondary wound closure.

To describe the quality of life in patients receiving a tertiary wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk class II, class III, class IV abdominal wounds
* Undergoing laparotomy for gynecologic related disorders
* Patients undergoing laparotomy for both benign and malignant diagnoses will be included in this study

Exclusion Criteria:

* Pregnancy
* Allergy to triclosan
* Patients undergoing HIPEC

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Percentage Comparisons of Tertiary Wound Closure Versus Historical Controls Postoperative Day 30 | 30 days after tertiary wound closure
  The percent of wound closure that occurs postoperative day #30 after tertiary wound closure as compared to historical controls receiving a secondary wound closure.

SECONDARY OUTCOMES:
Proportions of Tertiary Technique Versus Historical Controls | 30 days after tertiary wound closure
  The proportion of SSI using a tertiary closure technique compared to historical controls receiving a secondary would closure.
Length of Hospital Stay | Up to 3 months after surgery
  The length of stay as defined by the time from surgery to discharge as compared to historical controls receiving a secondary would closure.
Proportion of Patients Returning after Surgery | Up to 30 days after surgery
  The proportion of patients that return within 30 days of surgery.
Change of Quality of Life Questionnaire SF-36 | Up to 3 months after tertiary wound closure
  The quality of life in patients receiving a tertiary wound closure. The scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Kelly, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT03861065/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT03861065/ICF_000.pdf